CLINICAL TRIAL: NCT02773641
Title: Double Blind Placebo-controlled RCT of the Efficacy and Safety of Intramuscular Injections of Botulinum Toxin A as a Treatment for Provoked Vestibulodynia
Brief Title: Placebo-controlled RCT of Botulinum Toxin A as a Treatment for Provoked Vestibulodynia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nina Bohm-Starke, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BotA -KKDS2016, version 3
Record Dates: First submitted 2016-05-04; First posted 2016-05-16 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Type A (Active Comparator): 50 Allergan units (0.5 ml) injected in m bulbocavernosus twice with 3 months in between treatments
  Interventions: Drug: Botulinum Toxin Type A
- Sterile saline solution (Placebo Comparator): 0.5 ml of sterile saline injected in m bulbocavernosus twice with 3 months in between treatments
  Interventions: Drug: Sterile Saline Solution

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: Botox
  Arms: Botulinum Toxin Type A
Drug: Sterile Saline Solution
  Other Names: Sterile saline
  Arms: Sterile saline solution

SUMMARY:
Women with provoked vestibulodynia (PVD) suffer from severe dyspareunia and often present a hyperactivity of the pelvic floor muscles (PFM) which maintain the dyspareunia. The rationale for the study is that for women with PVD who don't succeed to restore the function of the PFM by physiotherapy, Botulinum Toxin A (BTA) could be an optional treatment by decreasing the high muscle tonus and thus possibly reduce the coital pain.

DETAILED DESCRIPTION:
Design and methodology General outline The study is an investigator- initiated phase III study to determine the effect of botulinum toxin A injections in the bulbocavernosus muscles in women with provoked vestibulodynia for reduction of the level of dyspareunia. The study will be a double blind, placebo-controlled RCT analyzed according to the intention to treat. The study will be carried out according the trial protocol, current regulations (LVFS 2011:19, ICH GCP) and to the latest version of the Helsinki declaration. Ethical approval from the Stockholm regional ethic committee will also be obtained before the study begins. No financial support from the manufacturer of the active drug is obtained.

Women with PVD, age 18-40 years, will be informed about the study by their gynecologist or via advertisement with information on how to contact the research nurse or the responsible gynecologists for more information. If the diagnosis of PVD needs to be clarified, a screening appointment will be scheduled.

It is estimated that the project will require 4 years for recruitment and treatment of all participants, follow-ups, data analyses and report of results.

During the recruitment, the patients with PVD will be asked to participate in an epigenetic study analyzing the grade of methylation of certain candidate genes associated to pain and anxiety before and after treatment and a "genome wide association study" with the aim to find possible genetic markers of PVD. If they accept, a venous blood sample will be taken during Visit 1 and Visit 5. These studies are otherwise separated from the RCT and have ethical approval. The blood samples will be registered in Stockholms Medicinska Biobank (registreringsnummer 941 hos IVO) and stored for later analyses at the research department of Dept. of Obstetrics and Gynecology, 182 88 Danderyd, Sweden.

Visit 1(recruitment and baseline) If the patient is willing to participate and fulfill inclusion and exclusion criteria she will sign informed consent in the presence of the gynecologist in charge of the injections of BTA or placebo.

Evaluation of psycho-sexual health and quality of life (QoL) The following validated (including the Swedish language) questionnaires will be filled in;

* Data on general and reproductive health including current medication and anti-conception method
* Female Sexual Function Index (FSFI)
* Female Sexual Distress Scale (FSDS)
* Quality of life (WHOQOL-BRIEF, Swedish version
* EQ-5
* PSS (perceived stress scale)
* Anxiety questionnaire (Spence, Swedish version).

Evaluation of coital pain/dyspareunia

* The level of dyspareunia the last month will be reported at baseline using VAS 0 (no pain) to 100 (worst pain imaginable)
* Functional measure of coital impairment (Never pain, Occasional or mild pain - not preventing intercourse, Moderate pain - sometimes preventing intercourse, Severe pain - most times preventing intercourse). In addition the
* Pain at insertion of a normal size tampon will also be reported according to VAS 0-100.

Vaginal pressure measurement Measurement of vaginal pressure will be performed by the use of a thin plastic catheter with a small pressure transducer at the top (4 mm), connected to a manometer. The catheter is placed in the vagina, 3 -4 cm from the vaginal opening. Vaginal resting pressure in mm Hg (VRP), pelvic floor muscle (PFM) strength, PFM endurance for 10s will be measured.

Venous blood sample of 20 ml to separate genetic studies

Randomization The research nurse will perform the randomization according to a computerized block-randomization and prepare sealed envelopes containing data of randomized treatment for each participant. She will also prepare a randomization list with name, personal number and randomization number that will be kept locked away in the research department.

Blinding and masking The research nurse who opens the randomization envelope will prepare the syringe with active drug or placebo according to the randomization number. The syringe will be marked with the patient's name, personal number and randomization number and left on a tray at an assigned place where it will be collected by the insertion provider (responsible investigator). Thus, a double blind procedure is obtained. Participation in the study and the patient's randomization number will be noted and kept in each patient's Clinical Research Format (CRF). Copies of the randomization envelopes will be kept locked away in the research department of the Dept. of Obstetrics and Gynecology, Danderyd Hospital. In case of emergency the individual envelopes can be obtained at all times and can then be accessed by all investigators involved in the study. Thereby the blinding of the study is not jeopardized in case of emergency.

Drug administration A total amount of 50 Allergan-units BTA, diluted in sterile NaCl solution 9 mg/ml to 0, 5 ml or 0, 5 ml of the sterile NaCl solution 9 mg/ml will be injected at two occasions (tree months apart) at 4 sites (2 at each side) in m. bulbocavernosus approximately 3-4 cm from the vaginal opening by EMG guidance and the use of an EMG needle (37mm x 27G, Natus Manufacturing Limited, Ireland).

Participants without a highly effective anti-conception method will undergo a pregnancy test before randomization and treatment. Highly anti-conception methods are defined as; combined hormonal method containing estrogen and progesterone (oral, intravaginal, transdermal), progesterone only (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tube occlusion, vasectomized partner, sexual abstinence.

In between visits, a web-based diary will be kept for reporting of adverse events, pain during sexual activity and the result of the tampon test performed once a week at home. The research nurse will send e-mails with the questionnaires to be filled in before each follow-up visit and check that all questionnaires have been completed. She will also remind the participants via e-mail to report adverse events and perform the tampon test as required.

Visit 2, 4-6 weeks after baseline

Evaluation of reported adverse events Vaginal pressure measurement

Visit 3, 12 weeks after baseline Evaluation of reported adverse events Questionnaires for psycho-sexual health and QoL - same as Visit 1

Coital pain and the tampon test (VAS 0-100) and functional measure of coital impairment Vaginal pressure measurement Pregnancy test of participants without highly effective anti-conception method The patients will be treated with the same treatment as they were randomized for at baseline (either 50 Allergan-units BTA (0.5 ml) or 0.5 ml placebo) injected in the same manner.

Visit 4, 16-18 weeks after baseline Evaluation of reported adverse events Vaginal pressure measurement

Visit 5, 24 weeks after baseline Evaluation of reported adverse events Questionnaires for psycho-sexual health and QoL - same as Visit 1

Coital pain and the tampon test (VAS 0-100) and functional measure of coital impairment

Vaginal pressure measurement Venous blood sample of 20 ml to separate genetic studies At this point patients will be offered, if needed, information on conventional treatment of PVD with exercises for desensitizing the vestibular mucosa and exercises pelvic floor muscles rehabilitation.

Visit 6, 12 months from baseline Questionnaires for psycho-sexual health and QoL - same as Visit 1

Coital pain and the tampon test (VAS 0-100), and functional measure of coital impairment

Vaginal pressure measurement

End of Trial

The trial is completed when the last patients has come for her Visit 6.

After the trial is completed, participants who have received placebo will be offered treatment with Botox injections, administered the same way as in the study, if the results show that Botox is more effective than placebo for PVD and that no serious adverse events have occurred during the trial. For the post-trial treatment, the patients have to pay for the medication. The treatment is otherwise free of charge. No other treatment for PVD is planned to be carried out and the participants will resume contact with their ordinary open care gynecologist if needed when the trial is completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* PVD defined as significant pain at vestibular contact and vaginal entry (VAS ≥ 6 at the tampon test or severe pain, preventing intercourse)
* Duration of symptoms of ≥ 3 months,
* 0-para,
* Patients who are willing to participate in the study after it has been explained orally and in writing will be included.

Exclusion Criteria:

* Vulvo-vaginal infection, dermatological conditions or other causes to dyspareunia
* Regular medication with analgesics
* Major psychiatric or medical disease
* Known allergy to any components of the active drug (Botox®) or medical disease contradictory to treatment with the active drug (Botox®) (peripheral motor neurological disease such as myasthenia gravis, amyotrophic lateral sclerosis or Lambert-Eaton syndrome and diabetes),
* Pregnancy - a pregnancy test will be taken before both treatments (Visit 1 and 3), unless the participants are using highly effective birth control methods that can achieve a failure rate of less than 1% per year, when used consistently and correctly. Such methods include;
* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* intrauterine device (IUD)
* intrauterine hormone-releasing system (IUS)
* bilateral tubal occlusion
* sexual abstinence (if refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the preferred and usual lifestyle of the subject.
* Pelvic floor deficiency with urine and or flatulence incontinence.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Self-reported dyspareunia measured by VAS | Baseline to 6 months after baseline
  VAS 0 (no pain) to 100 (worst pain imaginable)

SECONDARY OUTCOMES:
Pain at tampon insertion measured by VAS 0-100 | Baseline to 6 months after baseline
  VAS 0 (no pain) to 100 (worst pain imaginable)
Reduction of pelvic floor hyperactivity/tonus, | Baseline to 6 months after baseline
  Measured with a vaginal manometer
Quality of Life (questionnaires) | Baseline to 6 months after baseline
  Use of validated questionnaires
Psychosexual evaluations (questionnaires) | Baseline to 6 months after baseline
  Use of validated questionnaires
Registrations of adverse events | 1 year
  Adverse events will be registered according to the protocool

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bohm-Starke, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Dep. of Obstetrics and Gynecology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haraldson P, Muhlrad H, Heddini U, Nilsson K, Bohm-Starke N. Botulinum Toxin A for Provoked Vestibulodynia: 12 Months' Follow-up of a Randomized Controlled Trial. J Sex Med. 2022 Nov;19(11):1670-1679. doi: 10.1016/j.jsxm.2022.08.188. Epub 2022 Oct 26. PMID 36307361
- [Derived] Haraldson P, Muhlrad H, Heddini U, Nilsson K, Bohm-Starke N. Botulinum Toxin A as a Treatment for Provoked Vestibulodynia: A Randomized Controlled Trial. Obstet Gynecol. 2020 Sep;136(3):524-532. doi: 10.1097/AOG.0000000000004008. PMID 32769643